CLINICAL TRIAL: NCT01677390
Title: A Phase 1b, Open-label, Dose-escalation Study to Evaluate the Safety and Tolerability of SGN-75 in Combination With Everolimus in Patients With CD70-positive Metastatic Renal Cell Carcinoma
Brief Title: A Phase 1b Study of SGN-75 in Combination With Everolimus in Patients With Renal Cell Carcinoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGN75-002
Record Dates: First submitted 2012-08-23; First posted 2012-09-03 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2014-01

CONDITIONS: Renal Cell Carcinoma
Keywords: Antibody-Drug Conjugate; monomethylauristatin F; Carcinoma, Renal Cell; Antigens, CD70; Drug Therapy
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — SGN-75 antibody-drug conjugate; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): SGN-75, everolimus
  Interventions: Drug: SGN-75; Drug: everolimus

INTERVENTIONS:
Drug: SGN-75 — 1-2 mg/kg IV every 21 days
Drug: everolimus — 10 mg PO daily

SUMMARY:
This is a phase 1, open-label, dose-escalation clinical trial to evaluate the safety of SGN-75 in combination with everolimus in patients with CD70-positive metastatic renal cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of metastatic renal cell carcinoma with confirmed CD70 expression
* Previously treated with at least 1 tyrosine kinase inhibitor (TKI)
* Measurable disease
* Eastern Cooperative Oncology Group performance status 0 or 1
* Adequate lung and renal function

Exclusion Criteria:

* Prior treatment with anti-CD70-directed therapy
* Received more than one prior treatment with an mTOR inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events and laboratory abnormalities | Through 1 month post last dose

SECONDARY OUTCOMES:
Best clinical response according to RECIST Version 1.1 | Through 1 month post last dose
Progression-free survival | Until disease progression or start of new anticancer treatment, an expected average of 6 months
Overall survival | Until death or study closure, an expected average of 1 year
Blood concentrations of SGN-75 and metabolites | Cycle 1: pre-dose, 30 minutes, and 2, 4, 8, 24, 168, and 336 hours post dose start; pre-dose in subsequent cycles, and 1 month post last dose
Incidence of antitherapeutic antibodies | Pre-dose in most cycles and 1 month post last dose

CONTACTS AND LOCATIONS:
Overall Officials: Elaina Gartner, MD, Study Director — Seagen Inc.
Locations (8):
- United States (8):
  - Stanford Cancer Center, Stanford, California
  - Rocky Mountain Cancer Centers - Midtown, Denver, Colorado
  - Karmanos Cancer Institute / Wayne State University, Detroit, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - UNC Lineberger Comprehensive Cancer Center / University of North Carolina, Chapel Hill, North Carolina
  - Miriam Hospital, The, Providence, Rhode Island
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Seattle Cancer Care Alliance / University of Washington, Seattle, Washington